CLINICAL TRIAL: NCT06202677
Title: Effectiveness of a Self-guided Mobile Application in Improving Obsessive Compulsive Disorder Symptoms in Young Adults With Subclinical OCD - A Randomized Control Trial
Brief Title: Effectiveness of a Self-guided Mobile Application in Improving Obsessive Compulsive Disorder Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Intellect Pte. Ltd. (Industry)
Responsible Party: Principal Investigator, Dr Oliver Suendermann, Adjunct Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2023-444
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group: Obsessive Compulsive Disorder Program (Experimental): Participants will complete an 8-day self-guided programme on obsessive compulsive disorder delivered via a mobile phone application with daily exercises guided by cognitive-behavioural and exposure and response prevention principles.
  Interventions: Device: Self-guided program on obsessive compulsive disorder
- Control group (Active Comparator): Participants will complete an 8-day self-guided programme on cooperation delivered via a mobile phone application with daily exercises that differ from the intervention group in terms of content but are comparable in terms of duration.
  Interventions: Device: Self-guided program on cooperation

INTERVENTIONS:
Device: Self-guided program on obsessive compulsive disorder — This is an 8-day program that provides psychoeducational on what obsessions and compulsions are, and how to identify them. Subsequently, through a series of content learning and daily exercises that increase in difficulty, participants are guided to conduct exposure exercises while tolerating distress and refraining from compulsions. Participants are also guided to set goals and type down the specific content of their intrusive thoughts and compulsive behaviours to keep track of their progress. Each session of the program is estimated to be approximately 5 minutes.
  Arms: Experimental: Intervention group: Obsessive Compulsive Disorder Program
Device: Self-guided program on cooperation — This 8-day program on cooperation aims to improve participants' collaborative skills and interpersonal wellness through a series of content learning and practice exercises. The time and duration of this program is matched to the obsessive compulsive disorder program to ensure that participants spend a similar amount of time and effort across both the intervention and active control conditions.
  Arms: Control group

SUMMARY:
Obsessive Compulsive Disorder (OCD) is a significant mental health problem worldwide. OCD typically begins in young adulthood, and without adequate intervention, often takes a chronic course. Individuals with OCD may suffer impaired relationships, and ability to engage in leisure activities, study or work. Thus, prevention efforts are crucial to target OCD symptoms before they worsen.

The goal of this randomized-controlled trial (RCT) is to evaluate the effectiveness of a self-guided OCD program on a mobile phone application in young adults with subclinical OCD symptoms.

Hypothesis 1a: The intervention group will report significantly lower OCD symptoms (primary measure) at post-intervention and 1-month follow-up compared to the control group.

Hypothesis 1b. The intervention group will report significantly lower depression, anxiety and stress symptoms (secondary measure) at post-intervention and 1-month follow-up compared to the control group.

Hypothesis 2. Perfectionism will moderate the expected relationship between the OCD intervention and the reduction of scores on both primary and secondary measures, i.e. individuals with lower levels of perfectionism will benefit more from the OCD intervention than those with higher levels of perfectionism.

DETAILED DESCRIPTION:
Procedure:

Interested individuals will sign up for the study via an online survey link on the university's recruitment sites. They will first complete a pre-screening questionnaire on Qualtrics and be assessed on their eligibility based on the inclusion criteria (able to read and understand English, being a student from the National University of Singapore aged 18 to 30, and presenting with moderate subclinical OCD). Eligible participants read the Participation Information Sheet, and after providing informed consent, complete measures on depression, stress, anxiety, and perfectionism. They will also provide their demographic information (age, gender).

Next, participants are randomized to either the intervention or active control condition using simple randomization procedures and guided to download the mobile application on their mobile phone. Participants in the intervention group will undergo 8 days of the OCD learning program, while participants in the active waitlist control group will undergo 8 days of the cooperation learning program. Participation in each program is estimated to be about five minutes per day.

Upon completion of the 8-day program, participants will receive a survey link to complete measures on OCD, depression, anxiety, stress, and the App Engagement Scale. One month upon completion of the 8-day program, participants will be sent a survey link to the same survey, without the App Engagement Scale. They will also be briefed with an information sheet explaining the main purposes of the study. All participants will be given access to all well-being programs available on the app at the end of the study for their personal use. They will be reimbursed with either course credits or a small monetary fee for their participation in the study. Participants who chose to volunteer their participation will not be reimbursed.

Data screening:

Ineligible individuals, incomplete responses, long strings of identical responses, and outliers with data 3 standard deviations from the mean will be excluded from data analyses. Submissions with an overall response time of below 660s will be flagged.

Preliminary Analyses Statistical analyses will be done using SPSS Version 26.0. First, data will be visually inspected using scatterplots and histograms to examine the distribution of data and identify significant outliers. Analyses will be conducted with and without outliers to determine if outliers impact the results significantly. If results are significantly impacted by outliers, they will be will be replaced with the next closest non-outlying data point.

Data will be screened for normality and compliance with statistical assumptions. Independent t-tests and chi-square tests will examine the differences between the 2 conditions on all demographic and dependent variables.

Intent-to-treat analyses will be conducted to address missing data on questionnaires, by carrying forward the participants' last reported score. Missing data on the AES were accounted for using mean substitution.

Main analyses:

Assumptions for ANCOVA will first be conducted. For outcome measures where assumptions were violated, one-way ANOVA using difference scores. Thereafter, ANCOVA will be conducted to determine if changes in outcome measures at post-intervention and follow-up were significantly different between the two conditions. Baseline scores of the relevant outcome measure will be used as the covariate.

Moderation analyses:

Hayes PROCESS macro version 4.6 Model 1 will be used to conduct regression analysis between perfectionism and both primary and secondary measures. Confidence intervals will be set at 95% and bootstrapping samples = 5000.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 mild, subclinical OCD (OCI-R score of 0 to 20) Good command of the English language Owns a mobile phone for downloading the mobile application for use in the study's intervention Singaporean or Permanent Resident of Singapore

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
Change of obsessive compulsive disorder symptoms | Baseline, 8 days (completion of intervention), 4 weeks (follow-up)
  The Obsessive Compulsive Inventory - Revised (OCI-R; Foa et al., 2002) is used. The OCI-R is an 18-item self-report questionnaire which assesses OCD symptoms across 6 subscales: washing, checking, neutralising, obsessing, ordering, and hoarding. Each item is rated on a 5-point Likert scale with scores ranging from Not at all (0) to Extremely (4). The total score (ranging from 0-72) is the sum of all the items.

SECONDARY OUTCOMES:
Change of depression, anxiety and stress symptoms | Baseline, 8 days (completion of intervention), 4 weeks (follow-up)
  The Depression Anxiety Stress Scale-21 (DASS-21; Lovibond and Lovibond, 1995) is a set of three self-report scales assessing depression, anxiety and stress. Each subscale contains 7 items, totalling 21 items which are each rated on a 4-point Likert scale ranging from Did not apply to me at all (0) to Applied to me very much or most of the time (3). Three subscale scores and a total score can be computed by summing the items in each subscale.

OTHER OUTCOMES:
Perfectionism | Baseline
  The Frost Multidimensional Perfectionism Scale (FMPS; Frost et al.,1990) is a 35-item self-report scale which assesses perfectionism across 6 subscales: concern over mistakes (9 items), high personal standards (7 items), parental expectations (5 items), parental criticism (4 items), doubts about actions (4 items), and organisation (6 items). Each item is rated on a 5-point Likert scale ranging from Strongly disagree (1) to Strongly agree (5). The FMPS has demonstrated good internal consistency and convergent validity with other measures of perfectionism within non-clinical and clinical samples (Frost et al., 1990).
Engagement with the mobile application | 8 days (completion of intervention)
  The App Engagement Scale (AES; Bakker & Rikard, 2018) assesses app engagement. Each item is rated on a 5-point Likert scale with scores ranging from definitely disagree (1) to definitely agree (5). The total score (ranging from 1-35) is the sum of all the items.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Ph.D, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker D, Rickard N. Engagement in mobile phone app for self-monitoring of emotional wellbeing predicts changes in mental health: MoodPrism. J Affect Disord. 2018 Feb;227:432-442. doi: 10.1016/j.jad.2017.11.016. Epub 2017 Nov 9. PMID 29154165
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Foa EB, Huppert JD, Leiberg S, Langner R, Kichic R, Hajcak G, Salkovskis PM. The Obsessive-Compulsive Inventory: development and validation of a short version. Psychol Assess. 2002 Dec;14(4):485-96. PMID 12501574
- [Background] Frost, R. O., Marten, P., Lahart, C., & Rosenblate, R. The dimensions of perfectionism. Cognitive Therapy and Research. 1990; 14(5): 449-468.
- [Derived] Lee Yoon Li M, Lee Si Min S, Sundermann O. Efficacy of the mHealth App Intellect in Improving Subclinical Obsessive-Compulsive Disorder in University Students: Randomized Controlled Trial With a 4-Week Follow-Up. JMIR Mhealth Uhealth. 2024 Dec 16;12:e63316. doi: 10.2196/63316. PMID 39680884